CLINICAL TRIAL: NCT06109207
Title: The Safety and Feasibility of Neoadjuvant Camrelizumab With Dalpiciclib for the Treatment of Resectable Head and Neck Squamous Cell Carcinoma：A Phase 1 Trial
Brief Title: Neoadjuvant Camrelizumab With Dalpiciclib for Resectable Head and Neck Squamous Cell Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1551
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Squamous Cell Carcinoma; Neoadjuvant therapy; Immunotherapy; CDK4/6 inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab+Dalpiciclib(100mg) 3 patients (Experimental): Camrelizumab will be given at at a dose of 200 mg intravenously every three weeks on day 1 of a planned 21-day cycle, and two doses before surgery
  Dalpiciclib will be given at a dose of 100 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for two cycles.
  For dalpiciclib, there is 2 dose levels, 100mg qd and 150 mg qd, and if no patients experience DLT on 100mg level, 150mg level will be administered.
  Interventions: Drug: Camrelizumab; Drug: Dalpiciclib 100mg
- Camrelizumab+Dalpiciclib(150mg) 3 patients (Experimental): Camrelizumab will be given at at a dose of 200 mg intravenously every three weeks on day 1 of a planned 21-day cycle, and two doses before surgery
  Dalpiciclib will be given at a dose of 150 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for two cycles.
  For dalpiciclib, there is 2 dose levels, 100mg qd and 150 mg qd, and if no patients experience DLT on 100mg level, 150mg level will be administered.
  Interventions: Drug: Camrelizumab; Drug: Dalpiciclib 150mg

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab will be given at at a dose of 200 mg intravenously every three weeks on day 1 of a planned 21-day cycle, and two doses before surgery
Drug: Dalpiciclib 100mg — Dalpiciclib will be given at a dose of 100 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for two cycles.
  Arms: Camrelizumab+Dalpiciclib(100mg) 3 patients
Drug: Dalpiciclib 150mg — Dalpiciclib will be given at a dose of 150 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for two cycles.
  Arms: Camrelizumab+Dalpiciclib(150mg) 3 patients

SUMMARY:
The purpose of this study is to explore the safety and feasibility of anti-programmed cell death protein 1(PD-1) immunotherapy, Camrelizumab, combined with cyclin-dependent kinase 4/6 blockade, Dalpiciclib, as a new neoadjuvant treatment regimen for patients with resectable head and neck squamous cell carcinoma(HNSCC).

DETAILED DESCRIPTION:
Head and Neck Squamous Cell Carcinoma (HNSCC) is the most common malignancies of the head and neck, accounting for 90% of head and neck cancer. The 5-year survival rate under standard treatment is only 50%. 70%~80% of first diagnosed patients already developed into locally advanced status (stage II-Iva). In recent years, the use of neoadjuvant therapy (NAC) followed by surgery or radiotherapy has been advocated because of its higher probability of local/regional failure and distant metastasis after treatment. TPF (Docetaxel + Cisplatin + Fluorouracil) regimen is considered as the standard regimen of induced chemotherapy for head and neck squamous cell carcinoma (especially in laryngeal cancer), which can significantly reduce the patient's distant metastasis rate and prolong overall survival (OS). However, the therapeutic effect of neoadjuvant therapy on head and neck squamous cell carcinoma has reached a bottleneck. In recent years, PD-1 inhibitors have achieved significant effects in the field of tumor therapy and have been approved for the treatment of various tumors including recurrent metastatic head and neck tumors. There are also several prospective clinical research attempting to combine ICB with targeted therapeutic drugs for neoadjuvant therapy of HNSCC. The efficacy and safety results show potential synergy between these drugs.

Recent preclinical studies have shown that CDK4/6 inhibitors promote efficacy of PD-1/PD-L1 inhibitors through tumor antigen presentation enhancing, suppressed proliferation of regulatory T (Treg) cells, effector T- cell activation enhancing, and induction of T- cell memory. The previous study confirmed that CDK4/6 inhibitor combined with ICB can be administered safely in patients with recurrent or metastatic head and neck squamous cell carcinoma(HNSCC) and non-small cell lung carcinoma(NSCC).

In summary, the investigators designed this study to explore the safety and efficacy of anti-PD1 immunotherapy, Camrelizumab, combined with CDK4/6 inhibitor, dalpiciclib, as a new neoadjuvant treatment regimen for patients with resectable HNSCC. It will also provide new ideas, strategies, and experimental evidence for the development of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above.
* Patients with pathologically confirmed HNSCC (except for nasopharyngeal carcinoma) and meet the following conditions:

  * were newly diagnosed and without distant metastasis;
  * were deemed surgically resectable evaluated by a head and neck surgeon;
  * were willing to undergo surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate organ and bone marrow function: absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 80 g/L, platelets ≥ 80 × 10^9/L;ALT, AST and ALP < 2.5× upper limit of normal (ULN), total bilirubin ≤ 2×ULN;albumin≥ 2.8 g/dL；creatinine clearance ≥ 60 ml/min；INR≤ 1.5；APTT≤ 1.5×ULN
* Written informed consent.

Exclusion Criteria:

* History of other malignancies (except for the history of malignant tumors that have been cured and have not recurred within 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, in situ cervical cancer, and gastrointestinal mucosal cancer, etc.）
* Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
* Any history of allergic disease, or a sever hypersensitivity reaction to drugs, or allergy to the study drug components.
* Any of prior therapy with:anti-PD-1, anti-PD-L1/2, anti-CTLA-4 antibody, anti-EGFR antibody or EGFR-TKIs； antitumor vaccine; any active vaccine against an infectious disease within 4 weeks prior to the first dose or planned during the study period; major surgery or serious trauma within 4 weeks before the first dose; toxicity from prior antitumor therapy has not recovered to ≤ CTCAE Version 5.0 ·Grade 1 or the level specified by the inclusion/exclusion criteria.
* With serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart disease, supraventricular or ventricular arrhythmia, poorly controlled diabetes mellitus, poorly controlled hypertension, echocardiographic ejection fraction < 50%, etc.
* With interstitial pneumonitis, non-infectious pneumonitis, active pulmonary tuberculosis, or history of pulmonary tuberculosis infection that were not controlled by treatment.
* With hyperthyroidism, or organic thyroid disease.
* With active infection, or unexplained fever during the screening period or 48 hours before the first dose.
* With active hepatitis B or C, or known history of positive HIV test, or acquired immunodeficiency syndrome.
* History of a clear neurological or psychiatric disorder.
* History of drug abuse or alcohol abuse.
* Women who are pregnant or breastfeeding, or have a reproductive plan from the screening period to 3 months after the end of the study, or have sex without contraceptive measures, or are unwilling to take appropriate contraceptive measures.
* Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
* Any other factors that are not suitable for inclusion in this study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety of combination camrelizumab and dalpiciclib as assessed by number of participants who experience adverse events | Through the study completion, an average of 12 weeks
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Feasibility of combination camrelizumab and dalpiciclib as assessed by number of participants who experience adverse events | Through the study completion, an average of 12 weeks
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) as determined by number of participants with dose limiting toxicities (DLT) | Through the study completion, an average of 12 weeks
  Maximum tolerated dose will be determined by the maximum dose at which the least number of participants experience dose-limiting toxicity. The dose limiting toxicity is defined using the Common Terminology Criteria for Adverse Events (CTCAE).
Major Pathologic Response | Time of surgery
  Major Pathologic Response (MPR) was defined as fewer than 10% viable tumor cells.
Objective response rate (ORR) | Through the study completion, an average of 12 weeks
  Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of nivolumab and ipilimumab.
Progression free survival(PFS) | Up to 2 years
  Proportion of participants who achieve progression free survival post treatment
Overall survival (OS) | Up to 2 years
  Proportion of participants who achieve survival post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhou, MD.,PhD., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287
- [Background] Solomon B, Callejo A, Bar J, Berchem G, Bazhenova L, Saintigny P, Wunder F, Raynaud J, Girard N, Lee JJ, Sulaiman R, Prouse B, Bresson C, Ventura H, Magidi S, Rubin E, Young B, Onn A, Leyland-Jones B, Schilsky RL, Lazar V, Felip E, Kurzrock R. A WIN Consortium phase I study exploring avelumab, palbociclib, and axitinib in advanced non-small cell lung cancer. Cancer Med. 2022 Jul;11(14):2790-2800. doi: 10.1002/cam4.4635. Epub 2022 Mar 20. PMID 35307972
- [Background] Dennis MJ, Sacco AG, Qi Y, Bykowski J, Pittman E, Chen R, Messer K, Cohen EEW, Gold KA. A phase I study of avelumab, palbociclib, and cetuximab in patients with recurrent or metastatic head and neck squamous cell carcinoma. Oral Oncol. 2022 Dec;135:106219. doi: 10.1016/j.oraloncology.2022.106219. Epub 2022 Oct 21. PMID 36279618
- [Background] Mody MD, Rocco JW, Yom SS, Haddad RI, Saba NF. Head and neck cancer. Lancet. 2021 Dec 18;398(10318):2289-2299. doi: 10.1016/S0140-6736(21)01550-6. Epub 2021 Sep 22. PMID 34562395
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Saba NF, Steuer CE, Ekpenyong A, McCook-Veal A, Magliocca K, Patel M, Schmitt NC, Stokes W, Bates JE, Rudra S, Remick J, McDonald M, Abousaud M, Tan AC, Fadlullah MZH, Chaudhary R, Muzaffar J, Kirtane K, Liu Y, Chen GZ, Shin DM, Teng Y, Chung CH. Pembrolizumab and cabozantinib in recurrent metastatic head and neck squamous cell carcinoma: a phase 2 trial. Nat Med. 2023 Apr;29(4):880-887. doi: 10.1038/s41591-023-02275-x. Epub 2023 Apr 3. PMID 37012550
- [Background] Ju WT, Xia RH, Zhu DW, Dou SJ, Zhu GP, Dong MJ, Wang LZ, Sun Q, Zhao TC, Zhou ZH, Liang SY, Huang YY, Tang Y, Wu SC, Xia J, Chen SQ, Bai YZ, Li J, Zhu Q, Zhong LP. A pilot study of neoadjuvant combination of anti-PD-1 camrelizumab and VEGFR2 inhibitor apatinib for locally advanced resectable oral squamous cell carcinoma. Nat Commun. 2022 Sep 14;13(1):5378. doi: 10.1038/s41467-022-33080-8. PMID 36104359